CLINICAL TRIAL: NCT00918710
Title: Impact of the Human Papillomavirus (HPV) Status in Carcinologic Prognosis of Oropharynx Squamous Cell Carcinoma.
Brief Title: Human Papillomavirus and Oropharynx Carcinoma
Acronym: Papillophar
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOM 08104
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-03

CONDITIONS: Oropharyngeal Neoplasms
Keywords: Squamous cell carcinoma of Oropharynx; Human papillomavirus.; Biological prognostic markers.
MeSH Terms: conditions — Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pieces of Oropharyngeal squamous cell carcinomas biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with oropharyngeal squamous cell carcinomas

SUMMARY:
High risk papillomavirus (HR-HPV) have an oncogenic role in Oropharyngeal squamous cell carcinomas (OP-SCC) in at least 25% of the cases and the prevalence is increasing. HPV+ might be more chemo and radio sensible with a better prognosis (disease-free survival (DFS) and overall survival (OS) as compared to HPV negative OP-SCC ; hypothesis : 2y DFS > 20% improvement). The principal objective is to determine the impact of the status of HR-HPV in the prognosis of the OP-SCC. The principal criteria is the 2-years DFS.

Secondary objective : virologic characteristics of HPV+ tumors.

DETAILED DESCRIPTION:
The study has no impact on the treatment of the observed population. The clinical study include TNM status, previous story of HPV infection, smoking and alcoholic habits, treatment and outcome during 5 years. The virologic study include : HPV type, E6-E7 viral charge of HPV16, viral DNA integration in the tumoral genome, HPV16 variants, expression of HPV 16, 18, 31, 45 coding oncoproteins E6-E7 mRNA. Moreover a serologic study will be done.

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell carcinoma of Oropharynx proven histologically
* All stages TNM
* informed consent
* No previous or simultaneous Head Neck cancer
* Age >18

Exclusion Criteria:

* Squamous cell carcinoma other than oropharynx
* 2nd synchronous SCC localization
* No consent
* age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with squamous cell carcinoma of oropharynx followed by the participating centers
Sampling Method: Non-Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
DFS at 2 years in HPV + and - tumors | at 2 years

SECONDARY OUTCOMES:
Overall survival | At 2 years
HPV status | At the inclusion
Overall survival | At 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean LACAU, PhD, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Tenon Hospital, APHP, Paris, France

REFERENCES:
- [Derived] Pretet JL, Dalstein V, Touze A, Beby-Defaux A, Soussan P, Jacquin E, Birembaut P, Clavel C, Mougin C, Rousseau A, Lacau Saint Guily J; Papillophar Study Group. High levels of HPV16-L1 antibody but not HPV16 DNA load or integration predict oropharyngeal patient outcome: The Papillophar study. Clin Exp Med. 2023 Feb;23(1):87-96. doi: 10.1007/s10238-022-00796-2. Epub 2022 Feb 23. PMID 35199231